CLINICAL TRIAL: NCT04036604
Title: Investigation of The Effect of Pelvic Floor Exercise Programme Related to Sexual Dysfunction, Incontinence, Physical Activity Level and Quality of Life in Elderly.
Brief Title: Investigation of The Effect of Pelvic Floor Exercise Programme in Elderly.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Mehmet Sakıncı, Assos.Prof., Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-KAEK-20
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Pelvic Floor Muscle Weakness; Urinary Incontinence in Old Age; Sexual Dysfunction; Quality of Life
Keywords: Pelvic floor exercise; Urinary incontinence; Sexual dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Urinary Incontinence | interventions — Exercise; Educational Status

STUDY DESIGN:
Intervention Model Description: 2 groups Study Group and Control Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of pelvic floor exercise (Experimental): Group of pelvic floor exercise include 47 elderly people which contains contraction and repetition of pelvic floor muscle exercises during twice a week for 8 weeks performed by an expert pelvic health physiotherapist.
  Interventions: Other: Exercise
- Group of pelvic floor education (No Intervention): Group of pelvic floor education include 47 elderly people which contains anatomy of pelvic floor and dysfunction during once a week for 8 weeks performed by an expert pelvic health physiotherapist.

INTERVENTIONS:
Other: Exercise — Pelvic floor exercise programme include repetition of pelvic floor muscle contraction during twice a week for 8 weeks performed by an expert pelvic health physiotherapist.
  Pelvic floor education programme include pelvic floor anatomy, information about pelvic floor dysfunction and behavioral changes.
  Other Names: Education
  Arms: Group of pelvic floor exercise

SUMMARY:
Alteration of hormonal structure and decreasing of muscle tissue with aging causes pelvic floor dysfunction. Over age of 65 so many factors such as decrease in volume of muscle tissue, decrease in the amount of estrogen / testosterone, and low level of physical activity cause problems such as incontinence, prolapse, constipation and sexual dysfunction The aim of this study is to investigate the effectiveness of pelvic floor exercise program on sexual dysfunction, incontinence, quality of life and physical activity level in elderly.

DETAILED DESCRIPTION:
Pelvic floor problems including prolapse, voiding and defecation dysfunction have been seen in approximately 37% of women aged 60-79 years and incontinence is the leading pelvic floor dysfunction. The International Incontinence Society (ICS)defines that all types of involuntarily urinary leakage as urinary incontinence. The incidence of urinary incontinence is 26.6% in women aged 65-74 and 41.8% in patients aged 75 and over. Sexual dysfunction is also frequently encountered problem in pelvic floor disorders in people older than 65 years. The aim of this study is to investigate the effectiveness of pelvic floor exercise program on sexual dysfunction, incontinence, quality of life and physical activity level in elderly. Pelvic floor exercises programme contains different contractions of pelvic floor muscle. Each exercises have slow and fast twitch muscle exercise contraction.

ELIGIBILITY:
Inclusion Criteria:

To be aged over 65 To attend all exercise class Not to be communication problem

Exclusion Criteria:

To have neurogenic bladder To have metastatic prostate or ovary cancer To have enfection in urinary tractus To have pelvic organs malign diseases

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-06-02 (Actual)

PRIMARY OUTCOMES:
Female Sexual Dysfunction Index | 8 weeks
  The FSFI is a brief questionnaire measure of sexual functioning in women. It was developed for the specific purpose of assessing domains of sexual functioning (e.g. sexual arousal, orgasm, satisfaction, pain) in clinical trials.
International Index of Erectile Function Questionnaire | 8 weeks
  The 15-question International Index of Erectile Function (IIEF) Questionnaire is a validated, multi- dimensional, self-administered investigation that has been found useful in the clinical assessment of erectile dysfunction and treatment outcomes in clinical trials.
International Consultation on Incontinence Questionnaire- Short Form (ICIQ-SF) | 8 weeks
  The ICIQ-UI Short Form is a brief and psychometrically robust patient-completed questionnaire for evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence in men and women in research and clinical practice across the world. It is scored on a scale from 0-21.

SECONDARY OUTCOMES:
SEAPI-QMM | 8 weeks
  The SEAPI incontinence questionnaire includes 5 data points that rate severity of specific urinary symptoms. The SEAPI-QMM Incontinence Classification System was developed in the early 1990s as a system that could quantify urinary incontinence and its impact without special equipment or time-consuming procedures.
Physical Activity Scale for the Elderly (PASE) | 8 weeks
  Physical Activity Scale for the Elderly (PASE) is a brief (5 minutes) and easily scored survey designed specifically to assess physical activity in epidemiological studies of persons age 65 years and older[6].
  The PASE score combines information on leisure, household and occupational activity[7]. The PASE assesses the types of activities typically chosen by older adults (walking, recreational activities, exercise, housework, yard work, and caring for others. It uses frequency, duration, and intensity level of activity over the previous week to assign a score, ranging from 0 to 793, with higher scores indicating greater physical activity. PASE was initially developed in early 90s to provide an instrument to investigate specifically older people with an age-specific physical activity questionnaire, filling what was an important need in epidemiological research at that time

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sakıncı, Assos.Prof., Study Chair — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We have used SPSS for participant data after interventions

REFERENCES:
- [Result] Engberg S, Sereika SM. Effectiveness of Pelvic Floor Muscle Training for Urinary Incontinence: Comparison Within and Between Nonhomebound and Homebound Older Adults. J Wound Ostomy Continence Nurs. 2016 May-Jun;43(3):291-300. doi: 10.1097/WON.0000000000000227. PMID 27163683
- [Result] Serati M, Braga A, Di Dedda MC, Sorice P, Peano E, Biroli A, Torella M, Cromi A, Uccella S, Salvatore S, Ghezzi F. Benefit of pelvic floor muscle therapy in improving sexual function in women with stress urinary incontinence: a pretest-posttest intervention study. J Sex Marital Ther. 2015;41(3):254-61. doi: 10.1080/0092623X.2014.889052. Epub 2014 Mar 20. PMID 24512197